CLINICAL TRIAL: NCT00170417
Title: Clinical and Health Economic Benefit of Non-Pharmacological Treatment of Chronic Insomnia in Primary Care
Brief Title: Clinical Benefit of CBT for Insomnia in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Organization: NHS Greater Clyde and Glasgow (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZH/4/Z
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2000-12

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behaviour Therapy

SUMMARY:
The purpose of this study is to evaluate using an RCT the potential benefits of CBT for insomnia in the community

ELIGIBILITY:
Inclusion Criteria:

* Adult years (18+), living at home
* Meets clinical/RDC criteria for chronic insomnia

Exclusion Criteria:

* Deteriorating health
* Untreated major mental disorder

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2000-12; Study Completion 2003-05

CONTACTS AND LOCATIONS:
Overall Officials: Colin A Espie, PhD, Principal Investigator — University of Glasgow
Locations (1):
- Primary Care NHS, Glasgow and Edinburgh, United Kingdom